CLINICAL TRIAL: NCT02242786
Title: Response Assessment for External Beam Radiation Therapy in Spinal Metastasis of Hepatocellular Carcinoma (HCC): Usefulness of Diffusion-Weighted Magnetic Resonance (MR) Imaging as A Functional Imaging
Brief Title: Diffusion-Weighted Magnetic Resonance Imaging
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jong Won Kwon, Assistant Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013-07-174-003
Record Dates: First submitted 2014-08-22; First posted 2014-09-17 (Estimated); Last update posted 2014-11-07 (Estimated); Status verified 2014-11

CONDITIONS: Hepatocellular Carcinoma; Spine Metastasis
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EBRT (Experimental)
  Interventions: Radiation: External beam radiation therapy

INTERVENTIONS:
Radiation: External beam radiation therapy

SUMMARY:
Recently, diffusion-weighted (DW) MR imaging has widened its application on various oncologic applications. Especially, it is expected the DW MRI could provide valuable information about early response evaluation after treatment using rapid apparent diffusion coefficient (ADC) value change. It has demonstrated potential usefulness in response evaluation in the liver tumors after treatments such as transarterial chemoembolization (TACE) and radiation therapy (RT). Furthermore, it is a functional imaging technique that does not require a contrast agent, it can be safely used in patients with renal insufficiency or other medical contraindications for contrast agents.

The optimal assessment of early response of RT could provide one of the most important information to prescribe patient and cancer specific RT dose. It might be also important in palliative RT of HCC bone metastasis which is related with painful aggressive mass formation.

This study is performed to evaluate the usefulness of DW MRI in early response evaluation after RT for HCC bone metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Hepatocellular carcinoma
* Spine metastasis
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 3
* 20 or older age
* informed consent
* consent to birth control during 6 months after treatment

Exclusion Criteria:

* less than 12 weeks of expected survival
* indication of emergency operation
* uncontrolled ascites or encephalopathy
* previous RT field lesion (within in 1 month)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
oral morphine equivalent doseresponse criteria | 3 months after RT completion
  Degree of pain will be assessed via Visual Analog Scale for Pain (VAS).

SECONDARY OUTCOMES:
Modified Response Evaluation Criteria in Solid Tumor | 3 months after RT completion
Time to local tumor progression | From RT start to the date up to 24 weeks
Overall survival | From RT start to the date up to 24 weeks
Quality of Life | 3 months after RT completion
  Quality of life will be assessed via European Organization for Research and Treatment (EORTC)- Quality of Life Questionnaire (QLQ)-C15-PAL.

CONTACTS AND LOCATIONS:
Overall Officials: Jong Won Park, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea